CLINICAL TRIAL: NCT05362487
Title: Switching COPD Patients From Spiriva® HandiHaler® Maintenance Therapy to Spiriva® Respimat®: a Non-Interventional Real-world clinicAl ouTcome assEssment: NIS PIRATE
Brief Title: Assessment of Health-related Quality of Life After Switching COPD Patients From a Dry Powder Inhaler to a Soft Mist Inhaler Remaining on the Same Inhalative Drug
Acronym: NIS PIRATE
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0549
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients switching from Spiriva® HandiHaler® to Spiriva® Respimat®
  Interventions: Device: Spiriva® Respimat®; Device: Spiriva® HandiHaler®; Drug: Tiotropium bromide

INTERVENTIONS:
Device: Spiriva® Respimat® — Spiriva® Respimat®
Device: Spiriva® HandiHaler® — Spiriva® HandiHaler®
Drug: Tiotropium bromide — Tiotropium bromide

SUMMARY:
The objective of this non-interventional, observational study is to assess whether changing Chronic Obstructive Pulmonary Disease (COPD) patients from a dry powder inhaler (HandiHaler®) to a soft mist inhaler (Respimat®), without changing the pharmacological compound, will lead to an improvement in Clinical COPD Questionnaire (CCQ) score and in the scores of the three subdomains of CCQ score: symptoms (4 items), functional state (4 items) and mental state (2 items) during a study period of approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 40 years of age at baseline visit
* Patients with confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Patients who have been on Spiriva® HandiHaler® for ≥ 6 weeks at baseline visit
* Patients for whom a switch from Spiriva® HandiHaler® to Spiriva® Respimat® was planned prior to study inclusion. If additional inhalative COPD drugs (AICDs) are used: AICD treatment must have been stable for at least 6 weeks before study inclusion
* Signed written informed consent form to participation

Exclusion Criteria:

* Patients who have contraindications to Spiriva® Respimat® according to the current prescribing information label/ summary of product characteristics (SmPC)
* Patients who have signs of a current, acute respiratory tract infection 2 weeks prior visit 1
* Patients for whom further follow-up will not be possible at the enrolling site during the planned observational period (of approximately 8 weeks)
* Patients with confirmed diagnosis of only asthma
* Patients who had > 1 moderate to severe exacerbation(s) within the last 6 weeks prior to study inclusion
* Patients who are pregnant or breastfeeding
* Patients participating in an ongoing interventional study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) planned to be switched according to the respective Summary of product characteristics (SmPC) and consenting to participate in the study are eligible. To avoid any selection bias, all eligible patients will be invited to participate in this study, in the order in which their eligibility is determined.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hosp. Baselland,Univ.Med.Dept,Liestal, Liestal, Switzerland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a national, multicenter, non-interventional, observational, cohort study based on newly collected data with an observational period of at least 8 weeks until switch or discontinuation of Spiriva® Respimat® treatment or up to 52 weeks after baseline visit whatever occurs first.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the study. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
  Out of 9 patients who were screened only 4 participated in the study.
Groups:
- Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®: This arm includes patients with confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD) who were switched from Spiriva® HandiHaler® which contains 18 microgram tiotropium powder for inhalation to Spiriva® Respimat® which contains 2.5 microgram tiotropium per puff inhalation solution. The recommended daily dose of Spiriva® Respimat® for adults is 5 micrograms of tiotropium, equivalent to inhaling 2 puffs from the Respimat® inhaler once daily at the same time of day.
Period: Overall Study
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Started (Performed Visit 1 (baseline)) | 4
Perform Visit 2 (8 Weeks) | 3
Completed | 0
Not Completed | 4
Not completed — Study was prematurely terminated as per Sponsor's decision | 4

BASELINE CHARACTERISTICS:
Population: Patients who fulfilled all the eligibility criteria and participated in the baseline visit of the study.
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Clinical COPD Questionnaire score at baseline [Mean (Standard Deviation); unit: score on a scale] | 3.6 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 0.2 Points Decrease in the Clinical COPD Questionnaire (CCQ) Score Between Baseline and Visit 2 in Patients With High CCQ Baseline Score (≥ 2)
Description: Number of participants with 0.2 points decrease in the Clinical COPD Questionnaire (CCQ) score between baseline and visit 2 in patients with high CCQ baseline score (≥ 2) is reported.
  The CCQ contains 10 questions about symptoms (items 1, 2, 5, 6 of the CCQ), functional status (CCQ-4, items 7, 8, 9 and 10 of the CCQ) and mental state (items 3, 4 of the CCQ). Each of the 10 CCQ questions is scored by the patient on a 7-point scale (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. CCQ score values can be interpreted as: acceptable (CCQ < 1); acceptable for moderate disease (1 ≤CCQ <2); instable-severe limited (2 ≤ CCQ < 3); very instable-very severe limited (CCQ ≥ 3).
Time Frame: Baseline and at Week 8.
Population: Patients who fulfilled all the eligibility criteria, participated at the baseline visit and had post-baseline data for the primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Number of Participants With 0.2 Points Decrease in the CCQ Score Between Baseline and Visit 2 in Patients Independently From CCQ Baseline Score
Description: Number of participants with 0.2 points decrease in the CCQ score between baseline and visit 2 in patients independently from CCQ baseline score is reported.
  The CCQ contains 10 questions about symptoms (items 1, 2, 5, 6 of the CCQ), functional status (CCQ-4, items 7, 8, 9 and 10 of the CCQ) and mental state (items 3, 4 of the CCQ). Each of the 10 CCQ questions is scored by the patient on a 7-point scale (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. CCQ score values can be interpreted as: acceptable (CCQ < 1); acceptable for moderate disease (1 ≤CCQ <2); instable-severe limited (2 ≤ CCQ < 3); very instable-very severe limited (CCQ ≥ 3).
Time Frame: Baseline and at Week 8.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Changes in Clinical Control: Mean Change in the CCQ Score and in the Scores of the 3 CCQ Subdomains Symptom, Mental State, and Functional State Domain, in All Patients Independently From CCQ Baseline Score
Description: The CCQ contains 10 questions about symptoms (items 1, 2, 5, 6 of the CCQ), functional status (CCQ-4, items 7, 8, 9 and 10 of the CCQ) and mental state (items 3, 4 of the CCQ). Each of the 10 CCQ questions is scored by the patient on a 7-point scale (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The symptom score is calculation of the sum of the 4 items (items 1, 2, 5, 6) divided by 4. The mental state score is a calculation of the sum of the 2 items (items 3, 4) divided by 2. The functional state score is a calculation of the sum of the 4 items (items 7, 8, 9, 10) divided by 4. The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. CCQ score values and the CCQ subdomains score values can be interpreted as: acceptable (CCQ < 1); acceptable for moderate disease (1 ≤CCQ <2); instable-severe limited (2 ≤ CCQ < 3);very instable-very severe limited (CCQ ≥ 3).
Time Frame: Baseline and at Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 3
Units on a scale
  Change in CCQ score | 1.0 (0.3)
  Change in CCQ symptom subdomain score | 1.3 (0.0)
  Change in CCQ mental state subdomain | 0.8 (1.4)
  Change in CCQ functional state subdomain | 0.8 (0.4)

4. Secondary Outcome: Changes in Clinical Control: Mean Change in the CCQ Score and in the Scores of the 3 CCQ Subdomains Symptom, Mental State, and Functional State Domain, in Patients With High CCQ Baseline Score (≥ 2)
Description: The CCQ contains 10 questions about symptoms (items 1, 2, 5, 6 of the CCQ), functional status (CCQ-4, items 7, 8, 9 and 10 of the CCQ) and mental state (items 3, 4 of the CCQ). Each of the 10 CCQ questions is scored by the patient on a 7-point scale (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The symptom score is calculation of the sum of the 4 items (items 1, 2, 5, 6) divided by 4. The mental state score is a calculation of the sum of the 2 items (items 3, 4) divided by 2. The functional state score is a calculation of the sum of the 4 items (items 7, 8, 9, 10) divided by 4. The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. CCQ score values and the CCQ subdomains score values can be interpreted as: acceptable (CCQ < 1); acceptable for moderate disease (1 ≤CCQ <2); instable-severe limited (2 ≤ CCQ < 3); very instable-very severe limited (CCQ ≥ 3).
Time Frame: Baseline and at Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 3
Units on a scale
  Change in CCQ score | 1.0 (0.3)
  Change in CCQ symptom subdomain score | 1.3 (0.0)
  Change in CCQ mental state subdomain | 0.8 (1.4)
  Change in CCQ functional state subdomain | 0.8 (0.4)

5. Secondary Outcome: Breathlessness of the Patients at Baseline and at Week 8
Description: This outcome was planned to be assessed using the Modified Medical Research Council (mMRC) Questionnaire for Assessing the Severity of Breathlessness which contains one question scored by the patient on a 5-point scale between 0 and 4, with higher scores indicating severe breathlessness.
Time Frame: At baseline and at Week 8.
Population: Data for this Outcome Measure were not collected from any of the patients who attended the baseline study visit or the study visit at Week 8.
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Breathlessness of the Patients From Baseline to Week 8
Description: as for outcome 5
Time Frame: At baseline and at Week 8.
Population: as for outcome 5
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 8 weeks.
Description: Patients who fulfilled all the eligibility criteria and participated in the baseline visit of the study.
Arm/Group | Patients Switching From Spiriva® HandiHaler® to Spiriva® Respimat®
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05362487/Prot_SAP_000.pdf